CLINICAL TRIAL: NCT05781854
Title: Dexmedetomidine for Programed Intermittent Epidural Boluses Versus Continuous Epidural Infusion for Labour Epidural Analgesia: A Randomized Controlled Double-blind Trial
Brief Title: Dexmedetomidine for Intermittent Epidural Boluses Versus Continuous Epidural Infusion for Labour Epidural Analgesia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Khaled ahmed gomaa, principal investigator , anesthesiology and ICU resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dexmedetomidine in normallabor
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Analgesia, Epidural; Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (PIEB-group) (Active Comparator): After the initial epidural loading dose of 10 ml, 30 patients will receive programmed intermittent epidural boluses (5 ml every 45 min with the first bolus 30 minutes after epidural initiation) + patient controlled epidural analgesia (PCEA) as 5 ml boluses with a 20-minute lockout period).
  Interventions: Drug: Epidural analgesia with bupivacaine and dexmedetomidine
- Group C (CEI-group) (Active Comparator): After the initial epidural loading dose of 10 ml, 30 patients will receive continuous epidural infusion (5 ml/h starting immediately after the loading dose) + patient controlled epidural analgesia (PCEA) as 5 ml boluses with a 20-minute lockout period).
  Interventions: Drug: Epidural analgesia with bupivacaine and dexmedetomidine

INTERVENTIONS:
Drug: Epidural analgesia with bupivacaine and dexmedetomidine — Epidural analgesia with bupivacaine and dexmedetomidine

SUMMARY:
The aim of this study is to compare two modes of labour epidural analgesia:

programmed intermittent epidural boluses (PIEB) versus continuous epidural infusion (CEI), with patient controlled epidural analgesia (PCEA), using dexmedetomidine in addition to low-dose bupivacaine and through measuring the total volume of local anesthetic received through patient controlled epidural analgesia per hour

DETAILED DESCRIPTION:
Labour although varies with the individual may be the most painful experience, any women may ever encounter. Concerns about pain in labour are as old as mankind. Pain can make patients feel uncomfortable and become sleepless and agitated. Pain also stimulates the sympathetic nervous system, which causes increase in the heart rate, blood pressure, sweat production, endocrine hyper-function, and delays the patients' prognosis. Labor pain often causes a strong stress response. Several inhalation and parenteral anesthetics, sedatives, tranquilizers, and analgesics have been used for pain relief during labor, while over the last decade, lumbar epidural analgesia has greatly increased. The ideal labor analgesia should be based on maternal and child safety and should have a fast-acting good analgesic effect and less adverse reaction. Different adjuvants such as opioids and α2-adrenergic agonists were added to local anesthetics to improve the quality of intraoperative and postoperative analgesia. Dexmedetomidine is a highly selective 2-adrenergic agonist which has been used as pre-medication and as an adjuvant to general anesthesia . Dexmedetomidine have several beneficial actions during perioperative period. It decreases the sympathetic tone with attenuation of the neuroendocrine and hemodynamic response to anesthesia and surgery, reduce anesthetic and opioid requirement, cause sedation and analgesia. Dexmedetomidine was used to enhance the analgesic property of local anesthetics like lidocaine, bupivacaine and ropivacaine. The mechanism by which intrathecal alpha 2-adrenergic agonists prolong the motor and sensory block of local anesthetics is not clear. It may be an additive or synergistic effect secondary to the different mechanisms of action of local anesthetic and alpha 2-adrenergic agonist. Maintenance of epidural analgesia involved intermittent provider , administered boluses, patient-controlled epidural analgesia, and continuous epidural infusions with or without patient-controlled epidural analgesia. Continuous epidural infusion is the standard application setting for epidural infusion, highly effective, and provides consistent analgesia. however, is associated with greater local anesthetic consumption . A newer approach to maintenance of labor epidural analgesia involves the administration of programmed intermittent epidural boluses with patient-controlled epidural analgesia dosing for breakthrough pain. Earlier studies have suggested that programmed intermittent epidural boluses may be superior to continuous epidural infusion for labor analgesia and may be associated with a reduction in local anesthetic requirement, decreased motor blockade, lower risk of instrumental deliveries, and improved patient satisfaction. This may be related to increased pressure generated during automated boluses, resulting in improved distribution of the local anesthetic in the epidural space .

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 45 years
* Scheduled for normal vaginal delivery
* ASA physical status ӀI-IӀӀ.
* Singleton non-complicated pregnancy.
* At least 36 weak of gestation.
* Vertex presentation.

Exclusion Criteria:

* Patient refusal to epidural analgesia.
* History of cardiac, liver, or kidney diseases.
* History of allergy to amide local anesthetics or study medications.
* Any neurological problem.
* History of chronic opioid analgesic use.
* Any contraindication of regional anesthesia.
* Evidence of intrauterine growth restriction or fetal compromise.
* Failed or unsatisfactory analgesic block.
* Body mass index ≥40 kg/m2

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
total volume of local anesthetic | 24 hour
  total volume of local anesthetic received through patient controlled epidural analgesia per hour

SECONDARY OUTCOMES:
Ramsay sedation scale | 24 hour
  Completely awake or asleep and not responsive to any stimulus
Heart rate | 24 hour
  Beat per minute
Blood Pressure | 24 hour
  mmHg
Likert scale for satisfaction | 24 hour
  very satisfied or very dissatisfied
Bromage score for motor block | 24 hour
  free movement of legs and feet or unable to move legs and feet

CONTACTS AND LOCATIONS:
Overall Officials: Zein El-Abden Zareh Hassan, Professor, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Ebirim, L.N., Buowari, O.Y., Ghosh, S. Physical and Psychological Aspects of Pain in Obstetrics. In: Ghosh, S., editor. Pain in Perspective [Internet]. London: IntechOpen; 2012 [cited 2022 Oct 18]. Available from: https://www.intechopen.com/chapters/40395 doi: 10.5772/53923
- [Background] Fortescue C, Wee MYK. Analgesia in labour: non-regional techniques. Continuing Education in Anaesthesia, Critical Care, and Pain. 2005; 5(1): 219-223.
- [Background] Paramasivan A, Lopez-Olivo MA, Foong TW, Tan YW, Yap APA. Intrathecal dexmedetomidine and postoperative pain: A systematic review and meta-analysis of randomized controlled trials. Eur J Pain. 2020 Aug;24(7):1215-1227. doi: 10.1002/ejp.1575. Epub 2020 May 22. PMID 32333825
- [Background] Verghese T, Dixit N, John L, et al. Effect of intravenous dexmedetomidine on duration of spinal anaesthesia with hyperbaric bupivacaine - A comparative study. Indian J Clin Anaesth. 2019;6(1):97-101
- [Background] Mostafa MF, Herdan R, Fathy GM, Hassan ZEAZ, Galal H, Talaat A, Ibrahim AK. Intrathecal dexmedetomidine versus magnesium sulphate for postoperative analgesia and stress response after caesarean delivery; randomized controlled double-blind study. Eur J Pain. 2020 Jan;24(1):182-191. doi: 10.1002/ejp.1476. Epub 2019 Sep 12. PMID 31461801
- [Background] Martin E, Ramsay G, Mantz J, Sum-Ping ST. The role of the alpha2-adrenoceptor agonist dexmedetomidine in postsurgical sedation in the intensive care unit. J Intensive Care Med. 2003 Jan-Feb;18(1):29-41. doi: 10.1177/0885066602239122. PMID 15189665
- [Background] Gertler R, Brown HC, Mitchell DH, Silvius EN. Dexmedetomidine: a novel sedative-analgesic agent. Proc (Bayl Univ Med Cent). 2001 Jan;14(1):13-21. doi: 10.1080/08998280.2001.11927725. PMID 16369581
- [Background] Werdehausen R, Fazeli S, Braun S, Hermanns H, Essmann F, Hollmann MW, Bauer I, Stevens MF. Apoptosis induction by different local anaesthetics in a neuroblastoma cell line. Br J Anaesth. 2009 Nov;103(5):711-8. doi: 10.1093/bja/aep236. Epub 2009 Aug 22. PMID 19700777
- [Background] Fairbanks CA, Wilcox GL. Spinal antinociceptive synergism between morphine and clonidine persists in mice made acutely or chronically tolerant to morphine. J Pharmacol Exp Ther. 1999 Mar;288(3):1107-16. PMID 10027848
- [Background] Sng BL, Sia ATH. Maintenance of epidural labour analgesia: The old, the new and the future. Best Pract Res Clin Anaesthesiol. 2017 Mar;31(1):15-22. doi: 10.1016/j.bpa.2017.01.002. Epub 2017 Jan 12. PMID 28625301
- [Background] Ojo OA, Mehdiratta JE, Gamez BH, Hunting J, Habib AS. Comparison of Programmed Intermittent Epidural Boluses With Continuous Epidural Infusion for the Maintenance of Labor Analgesia: A Randomized, Controlled, Double-Blind Study. Anesth Analg. 2020 Feb;130(2):426-435. doi: 10.1213/ANE.0000000000004104. PMID 30882524
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] El Fawal, S., El Kabarity, R., Ahmed, N., Abd-El-Tawab, S. (2022). Effect of Epidural Dexmedetomidine vs Nalbuphine for Labor Analgesia. A randomized clinical trial. Egyptian J Anesthesia: 38 (1); 373382